CLINICAL TRIAL: NCT05127928
Title: Antioxidants Vitamins and Muscle Damage
Acronym: Antioxidant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, María Martínez Ferrán, PhD student, principal investigator, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIPI/20/209-part2
Record Dates: First submitted 2021-06-15; First posted 2021-11-19 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Oxidative Stress
Keywords: antioxidant vitamins; oxidative damage
MeSH Terms: interventions — Vitamin E; Ascorbic Acid; Tocopherols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplementation (Experimental): Vitamin C and Vitamin E before exercise
  Interventions: Dietary Supplement: Dietary Supplement: Vitamin C and vitamin E
- Placebo (Placebo Comparator): Placebo before exercise
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Vitamin C and vitamin E — Antioxidant supplementation
  Other Names: Ascorbic acid and tocopherol
  Arms: Supplementation
Dietary Supplement: Placebo — Placebo administration
  Arms: Placebo

SUMMARY:
Determine if acute supplementation with antioxidant vitamins (vitamin C and vitamin E) influences the muscle damage and fatigue caused after an acute session of eccentric training.

DETAILED DESCRIPTION:
A randomized, single-blind, placebo-control parallel trial will be conducted. In a previous session volunteers will be interviewed to determine if they meet the inclusion criteria.

Participants should avoid ingesting of foods that contain high amounts of antioxidant compounds: more than two juices of fruits, more than four cups of coffee or tea. Juices with high antioxidant content should be avoided. Alcoholic beverages should also be avoided. Participants will be divided in to groups and will performance one resistance exercise sessions. Prior to exercise, one group will intake supplementation VitC (1000 mg) + VitE (235 mg) and the other supplementation with placebo.

The following sequence will be performed in each session: 1) baseline assessment (analysis of the composition body, blood draw and parameters of performance) prior to exercise session ; 2) administration of vitamin or placebo supplementation 2 hours before exercise session ; 3) post-exercise assessments (blood biomarkers and performance parameters) immediately after the session and after 24 hours. DOMS will also be assessed 48 h and 72 h after training. The training session implemented will be designed by a Sport Scientific

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Physically active

Exclusion Criteria:

* Injuries
* Supplementation or drugs
* Smokers

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-06 (Actual)

PRIMARY OUTCOMES:
Percentage of body fat and muscle mass | Prior to the intervention
  Determination of body composition using skinfolds measurements
DOMS | 0 hours post exercise
  Delayed onset muscle soreness. This outcome will be measure with a 10-point visual analogic scale (0= no pain; 10 = worst possible pain)
DOMS | 24 hours post exercise
  Delayed onset muscle soreness. This outcome will be measure with a 10-point visual analogic scale (0= no pain; 10 = worst possible pain)
Blood malondialdehyde (MDA) | 2 hours prior to exercise
  MDA will be analyzed from a blood sample
Blood creatine quinase (CK) | 2 hours prior to exercise
  CK will be analyzed from a blood sample
Blood malondialdehyde (MDA) | Inmediatly after exercise
  MDA will be analyzed from a blood sample
Blood malondialdehyde (MDA) | 24 hours after exercise
  MDA will be analyzed from a blood sample
Blood creatine quinase (CK) | 24 hours after exercise
  CK will be analyzed from a blood sample
Jump height in a Counter Movement Jump | 2 hours prior to exercise
  Jump height (cm) in a counter movement jump measured with Octojump Platform
Jump height in a Counter Movement Jump | Inmediatly after exercise
  Jump height (cm) in a counter movement jump measured with Octojump Platform
Jump height in a Counter Movement Jump | 24 h after exercise
  Jump height (cm) in a counter movement jump measured with Octojump Platform
Jump Height in a Squat Jump | 24 h after exercise
  Jump Height (cm) in a Squat Jump measured with Octojump Platform
Jump Height in a Squat Jump | Inmediately after exercise
  Jump Height (cm) in a Squat Jump measured with Octojump Platform
Jump Height in a squat Jump | 2 hours prior to exercise
  Jump height (cm) in a squat jump with Octojump Platform measured with Octojump Platform
Jump Height in a Drop Jump | 2 hours prior to exercise
  Jump height (cm) was measured in different drop jumps with Octojump Platform
Jump Height in a Drop Jump | Inmediately after exercise
  Jump height (cm) was measured in different drop jumps with Octojump Platform
Contact time in a Drop Jump | Inmediately after exercise
  Contact time (s)measured in different drop jumps with Octojump Platform
Jump Height in a Drop Jump | Inmediately after exercise
  Jump height (cm) measured in different drop jumps with Octojump Platform
Contact time in a Drop Jump | 24 hours after exercise
  Contact time (s) measured in different drop jumps with Octojump Platform
Jump Height in a Drop Jump | 24 hours after exercise
  Jump height (cm) measured in different drop jumps with Octojump Platform
Contact time in a Drop Jump | Inmediately after exercise
  Capillary blood lactate evaluated with Lactate Pro 2
Concentration of blood lactate | 2 hours before exercise
  Capillary blood lactate with Lactate Pro 2

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No